CLINICAL TRIAL: NCT00831766
Title: A Phase 1/2 Study of Sequential Idarubicin + Cytarabine, Followed by Lenalidomide, in Patients With Myelodysplastic Syndrome (RAEB-2) or With Previously Untreated Acute Myeloid Leukemia
Brief Title: Idarubicin + Cytarabine and Lenalidomide in Patients With Myelodysplastic Syndrome (MDS), Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15625; RV-AML/MDS-PI-0269 (Other: Celgene)
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: Hematopoietic; Myeloid and Monocytic Leukemia; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute | interventions — Idarubicin; Antineoplastic Agents; Cytarabine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I: Dose Escalation (Experimental): Induction: A dose escalation plan for induction therapy using a standard 3x3 design with dose escalation of Lenalidomide only, to determine maximum tolerated dose (MTD). Idarubicin and cytarabine doses will be fixed.
  Idarubicin: 12 mg/m^2.
  Cytarabine: 200 mg/m^2.
  Lenalidomide: According to dose escalation levels. Level 1: 5 mg/d; Level 2: 10 mg/d; Level 3: 15 mg/d; Level 4: 20 mg/d; Level 5: 25 mg/d.
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Lenalidomide (Revlimid®)
- Phase II: Treatment at MTD (Experimental): Idarubicin: 12 mg/m^2.
  Cytarabine: 200 mg/m^2.
  Lenalidomide: Maximum Tolerated Dose (MTD).
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Lenalidomide (Revlimid®)

INTERVENTIONS:
Drug: Idarubicin — Intravenous infusion of Idarubicin as outlined in Phase I and Phase II Treatment Arms.
  Other Names: Antineoplastic Agent
Drug: Cytarabine — Intravenous infusion of Idarubicin as outlined in Phase I and Phase II Treatment Arms.
  Other Names: Antineoplastic Agent
Drug: Lenalidomide (Revlimid®) — Lenalidomide as outlined in Phase I and Phase II Treatment Arms.
  Other Names: Revlimid®

SUMMARY:
The purpose of this study is to:

* Test the safety of the research study drug, lenalidomide, when given with Idarubicin and Cytarabine
* See how many respond to combination treatment with lenalidomide, Idarubicin and Cytarabine
* See how long people respond to this combination therapy
* See how long people live after being treated with this combination of drugs

DETAILED DESCRIPTION:
All three drugs are FDA approved to treat patients in the United States of America. Idarubicin and Cytarabine combination therapy is a standard treatment for patients with acute myeloid leukemia (AML). Lenalidomide is FDA approved to retreat patients with Multiple Myeloma or Myelodysplastic syndrome with a specific change in their DNA. Loss of a specific part of DNA is also seen in some patients with AML.

This is a phase 1/2, dose-escalation trial of Lenalidomide given in combination with idarubicin + cytarabine. During phase 1, we will enroll patients with AML involving del 5q31; 2) patients with MDS RAEB-2 associated with monosomy 5 or segmental deletion involving 5q31, either alone or with additional cytogenetic abnormalities, and 3) older patients with any type of karyotypic profile in whom an effective and reliable standard of care remains to be developed. All 3 groups of patients define a population of patients with very poor prognoses. Dose escalation of lenalidomide will use a standard 3x3 design. Dose escalation of Lenalidomide only will take place, while the doses of idarubicin and cytarabine will be constant. This trial will have an induction component, consolidation component, and maintenance component. Overall safety and MTD will be determined from the induction phase only.

During phase 2, we will enroll only patients with AML age ≥ 60 years. During phase 2, the efficacy of this combination of Lenalidomide + idarubicin + cytarabine, at the maximum tolerated dose (MTD) for Lenalidomide (determined during phase 1), will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Disease-specific criteria (Phase I):

  * Previously untreated Acute Myeloid Leukemia (AML), associated with monosomy 5 or segmental deletion involving 5q31, either alone or with additional cytogenetic abnormalities
  * Previously untreated AML (age ≥ 60 years)
  * Myelodysplastic Syndrome, Refractory Anemia with Excess Blasts-2 (MDS,RAEB-2, 10-19% blasts in the bone marrow) associated with monosomy 5 or segmental deletion involving 5q31, either alone or with additional cytogenetic abnormalities
  * For MDS, patients must have had progression with or failed response to front-line therapy with a nucleoside analogue (azacitidine, decitabine).
* Disease Specific Criteria (Phase II)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Laboratory test results within these ranges:

  * Serum creatinine ≤ 2.0 mg/dL
  * Total bilirubin ≤ 1.5 mg/dL (Gilbert's syndrome excluded)
  * Aspartic transaminase (AST) and Alanine transaminase (ALT) ≤ 2 x upper limit of normal (ULN)
* Disease free of prior malignancies for ≥ 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide. For FCBP who have a medical need to proceed with therapy immediately, the pregnancy test that would normally be done 10-14 days prior to initiation of lenalidomide may be done as late as 7 days prior to initiation of lenalidomide. Both this test and the pregnancy testing done within 24 hours prior to initiation of lenalidomide must be negative. FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex* condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. *For patients who have latex allergies or whose partner(s) have latex allergies, alternatives will be discussed.
* Must be able to swallow capsules and no evidence of gastrointestinal (GI) tract abnormality that would alter absorption of oral medications
* Understand and voluntarily sign an informed consent form
* Life expectancy >3 months
* All study patients must be registered into the mandatory RevAssist® program and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by RevAssist) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Unwilling or unable to participate with Food and Drug Administration (FDA) mandated birth control and pregnancy guidelines
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* The development of erythema nodosum, if characterized by a desquamating rash, while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* AML with cytogenetics including t(15;17), t(8;21), or inv(16)
* White blood count (WBC) count ≥ 50,000 on hydroxyurea therapy
* Previous history of induction chemotherapy for AML or allogeneic stem cell transplant
* Predicted inability to tolerate standard induction chemotherapy with idarubicin and cytarabine
* History of spontaneous thromboembolic event requiring use of anticoagulation with warfarin (coumadin) or low molecular-weight heparin within 3 years
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-06-25 (Actual); Primary Completion 2015-02-17 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lancet, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center and Cleveland Clinic between June 2009 and March 2014.
Groups:
- Phase I: Dose Escalation: Induction: A dose escalation plan for induction therapy using a standard 3x3 design with dose escalation of Lenalidomide only, to determine maximum tolerated dose (MTD). Idarubicin and cytarabine doses will be fixed.
  Idarubicin: 12 mg/m^2.
  Cytarabine: 200 mg/m^2.
  Lenalidomide: According to dose escalation levels. Level 1: 5 mg/d; Level 2: 10 mg/d; Level 3: 15 mg/d; Level 4: 20 mg/d; Level 5: 25 mg/d.
  Idarubicin: Intravenous infusion of Idarubicin as outlined in Phase I and Phase II Treatment Arms.
  Cytarabine: Intravenous infusion of Idarubicin as outlined in Phase I and Phase II Treatment Arms.
  Lenalidomide (Revlimid®): Lenalidomide as outlined in Phase I and Phase II Treatment Arms.
- Phase II: Treatment at MTD: Idarubicin: 12 mg/m^2.
  Cytarabine: 200 mg/m^2.
  Lenalidomide: Maximum Tolerated Dose (MTD).
  Idarubicin: Intravenous infusion of Idarubicin as outlined in Phase I and Phase II Treatment Arms.
  Cytarabine: Intravenous infusion of Idarubicin as outlined in Phase I and Phase II Treatment Arms.
  Lenalidomide (Revlimid®): Lenalidomide as outlined in Phase I and Phase II Treatment Arms.
Period: Overall Study
Arm/Group | Phase I: Dose Escalation | Phase II: Treatment at MTD
Started | 23 | 28
Completed | 23 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled, according to study phase. Outcome measure groups may vary depending on the analysis required.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Escalation | Phase II: Treatment at MTD | Total
Number analyzed (Participants) | 23 | 28 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 15 | 23 | 38
Age, Continuous [Mean (Full Range); unit: years] | 65 [35 to 79] | 70 [60 to 82] | 67.7 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 18 | 15 | 33
Region of Enrollment [Number; unit: participants]
  United States | 23 | 28 | 51

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose
Description: For the Phase I component, no formal statistical analysis was planned. The primary endpoint is to determine the maximum tolerated dose (MTD) and recommended Phase II dose of lenalidomide given in combination with standard idarubicin + cytarabine induction therapy.
Time Frame: 18 months
Population: Phase I participants.
Measure: Number; unit: mg/day
Groups:
- Phase I Participants: Dose escalation group.
Arm/Group | Phase I Participants
Number analyzed (Participants) | 23
mg/day | 20

2. Primary Outcome: Phase II: Complete Response Rate of Participants Treated at Maximum Tolerated Dose (MTD)
Description: Percentage of participants achieving CR/CRi. Complete Response (CR) plus Complete Response with Incomplete Count Recovery (CRi) rates. Response rates (CR + CRi) of lenalidomide following idarubicin and cytarabine induction therapy in older patients with previously untreated AML. A CR designation requires that the patient achieve the morphologic leukemia-free state and have an absolute neutrophil count of more than 1,000/μL and platelets of 100,000/μL. CRi: After chemotherapy, patients fulfill all of the criteria for CR except for residual neutropenia (1,000/μL) or thrombocytopenia (100,000/μL).
Time Frame: 24 months
Population: All participants treated at MTD
Measure: Number; unit: percentage of participants
Groups:
- All Participants Treated at MTD: All participants, regardless of Phase who were treated at the maximum tolerated dose (MTD).
Arm/Group | All Participants Treated at MTD
Number analyzed (Participants) | 39
percentage of participants | 54

3. Secondary Outcome: Rate of Lenalidomide Related Toxicity During Maintenance Therapy
Description: Rate of toxicities of lenalidomide as maintenance therapy according to the National Cancer Institute Common Toxicity Criteria (CTC) V3. Adverse Events: Possibly Related; Probably Related, or Definitely Related to study treatment. Events are categorized as Grade 1 or 2, or as Grade 3 or 4.
Time Frame: 24 months
Population: All Maintenance Phase participants.
Measure: Count of Participants; unit: Participants
Groups:
- Maintenance Phase Participants: All participants treated in the Maintenance Phase.
Arm/Group | Maintenance Phase Participants
Number analyzed (Participants) | 6
Participants
  Leukocytes (total WBC) - low - Grade 1 or 2 | 1
  Leukocytes (total WBC) - low - Grade 3 or 4 | 0
  ANC/AGC - Grade 1 or 2 | 0
  ANC/AGC - Grade 3 or 4 | 1
  Platelets - low - Grade 1 or 2 | 3
  Platelets - low - Grade 3 or 4 | 0
  Fatigue - Grade 1 or 2 | 1
  Fatigue - Grade 3 or 4 | 0
  Dry skin - Grade 1 or 2 | 1
  Dry skin - Grade 3 or 4 | 0
  Pruritus/itching - Grade 1 or 2 | 1
  Pruritus/itching - Grade 3 or 4 | 0
  Rash/desquamation - Grade 1 or 2 | 2
  Rash/desquamation - Grade 3 or 4 | 0
  Constipation - Grade 1 or 2 | 1
  Constipation - Grade 3 or 4 | 0
  Diarrhea - Grade 1 or 2 | 2
  Diarrhea - Grade 3 or 4 | 0
  Nausea - Grade 1 or 2 | 1
  Nausea - Grade 3 or 4 | 0
  Ulcer, GI - Anus - Grade 1 or 2 | 1
  Ulcer, GI - Anus - Grade 3 or 4 | 0
  Hemorrhage, GI - Rectum - Grade 1 or 2 | 1
  Hemorrhage, GI - Rectum - Grade 3 or 4 | 0
  Infection - Skin (cellulitis) Grade 1 or 2 | 1
  Infection - Skin (cellulitis) Grade 3 or 4 | 0
  AST, SGOT - Grade 1 of 2 | 2
  AST, SGOT - Grade 3 or 4 | 0
  Pain - Head/headache - Grade 1 or 2 | 1
  Pain - Head/headache - Grade 3 or 4 | 0

4. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival (PFS), defined as the time from study entry to disease progression, relapse, or death due to any cause, whichever is earlier, will be summarized with the Kaplan-Meier curve.
Time Frame: 24 months
Population: All participants treated at MTD.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants Treated at MTD
Number analyzed (Participants) | 39
months | 7.55 [5.53 to 10.53]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Overall Survival (OS), defined for those patients who have achieved CR or CRi as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier, to be analyzed similarly. Descriptive analysis was planned for this measure.
Time Frame: Up to 24 Months
Population: All participants treated at MTD
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants Treated at MTD
Number analyzed (Participants) | 39
months | 11.22 [7.61 to 13.74]

6. Other Pre Specified Outcome: Rate of Cytogenetic Remission Following Induction Therapy
Description: Rate of cytogenetic remission following induction therapy. Descriptive analysis was planned for this measure.
Time Frame: 24 Months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Median Relapse-Free Survival (RFS)
Description: Relapse-Free Survival (RFS), defined for those patients who have achieved CR or CRi as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier, will be analyzed similarly. Descriptive analysis was planned for this measure.
Time Frame: 24 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years, 8 months
Description: All Serious Adverse Events (SAEs) are reported, regardless of causality. All Other (not including Serious) Adverse Events (AEs) meeting 5% frequency threshold are reported, regardless of causality.
Groups:
- Phase I: Dose Escalation: Participants enrolled during Phase I.
- Phase II: Treatment at MTD: Participants enrolled during Phase II.
Arm/Group | Phase I: Dose Escalation | Phase II: Treatment at MTD
Serious Adverse Events (participants affected / at risk) | 5/23 | 13/28
Other Adverse Events (participants affected / at risk) | 22/23 | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Escalation (N=23) | Phase II: Treatment at MTD (N=28)
Neutrophils/granulocytes - low (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Platelets - low (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac Arrhythmia - Other, atrial fibrilation with rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmai - atrial fibirillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia) (General disorders) | 1 (1) | 1 (1)
Death - Disease progression NOS (General disorders) | 1 (1) | 0 (0)
Death - Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Mucositis/stomatitis - Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 9 (9)
Infection with Grade 3 or 4 neutrophils - abdomen, NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 0 (0) | 5 (5)
Infection with Grade 3 or 4 neutrophils - Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophnils - Gallbladder (cholecystitis) (Infections and infestations) | 0 (0) | 1 (1)
AST, SGOT - high (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Extremity, limb (General disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other, acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 Neutrophils - Urinary Tract (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Escalation (N=23) | Phase II: Treatment at MTD (N=28)
Diarrhea (Gastrointestinal disorders) | 19 (31) | 25 (41)
Nausea (Gastrointestinal disorders) | 12 (16) | 16 (33)
Constipation (Gastrointestinal disorders) | 7 (7) | 17 (19)
Anorexia (Gastrointestinal disorders) | 6 (7) | 16 (23)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 9 (11) | 13 (18)
Vomiting (Gastrointestinal disorders) | 7 (8) | 15 (17)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 11 (17)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 7 (7)
Gastrointestinal - Other, GERD (Gastrointestinal disorders) | 0 (0) | 3 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 5 (5)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (4) | 5 (11)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 5 (6)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 14 (25) | 19 (35)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 (6) | 14 (18)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (9)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Infections and infestations) | 14 (22) | 22 (39)
Infection with Grade 3 or 4 neutrophils - Lung (pneumonia) (Infections and infestations) | 9 (12) | 5 (5)
Infection with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 0 (0) | 9 (10)
Infection with Grade 3 or 4 neutrophils - Skin (cellulitis) (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 (1) | 3 (3)
Infection with Grade 3 or 4 neutrophils - Abdomen NOS (Infections and infestations) | 1 (1) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 2 (2) | 1 (2)
Infection with unknown ANC - Skin (cellulitis) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Infection with Grade 3 or 4 neutrophils - Anal/perianal (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Infection with Grade 3 or 4 neutrophils - Bladder (urinary) (Infections and infestations) | 0 (0) | 2 (2)
Infection with unknown ANC - Anal/perianal (Infections and infestations) | 0 (0) | 2 (2)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (1) | 2 (2)
Platelets - low (Blood and lymphatic system disorders) | 16 (22) | 17 (40)
Hemoglobin - low (Blood and lymphatic system disorders) | 9 (16) | 18 (31)
Neutrophils/granulocytes - low (Blood and lymphatic system disorders) | 10 (12) | 14 (30)
Leukocytes (total WBC) - low (Blood and lymphatic system disorders) | 2 (4) | 6 (16)
Pain - Abdomen NOS (General disorders) | 10 (13) | 7 (9)
Pain - Head/headache (General disorders) | 1 (1) | 11 (12)
Pain - Chest wall (General disorders) | 3 (3) | 7 (8)
Pain - back (General disorders) | 2 (2) | 6 (6)
Pain - Throat/pharynx/larynx (General disorders) | 2 (3) | 6 (7)
Pain - Chest/thorax NOS (General disorders) | 1 (1) | 5 (5)
Pain - Extremity-limb (General disorders) | 1 (2) | 2 (3)
Pain - Oral cavity (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 5 (6) | 14 (16)
Rigors/chills (General disorders) | 3 (4) | 13 (20)
Insomnia (General disorders) | 3 (3) | 10 (11)
Fever (in the absence of neutropenia) (General disorders) | 5 (6) | 14 (16)
Sweating (diaphoresis) (General disorders) | 1 (1) | 5 (6)
Weight loss (General disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 15 (19)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 13 (16)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Pulmonary/Upper Respiratory - Other, respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 8 (11) | 18 (29)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Lymphatics - Other, fluid retention (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
ALT, SGPT - high (Metabolism and nutrition disorders) | 5 (6) | 7 (12)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (4) | 7 (11)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (11) | 5 (5)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (5) | 6 (8)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (7) | 3 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (6) | 4 (8)
AST, SGOT - high (Metabolism and nutrition disorders) | 3 (4) | 6 (7)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6 (8) | 2 (4)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (12) | 1 (1)
Alkaline phosphatase - increased (Metabolism and nutrition disorders) | 3 (5) | 2 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Creatinine - high (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5) | 12 (17)
Mood alteration - Anxiety (Psychiatric disorders) | 4 (4) | 8 (8)
Confusion (Nervous system disorders) | 1 (2) | 4 (4)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 (0) | 6 (6)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 2 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2)
Mental status - Change (Psychiatric disorders) | 0 (0) | 4 (4)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (11)
Petechiae/purpura (hrmorrhage/bldding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Hemorrhage, G I- Oral cavity (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 3 (4) | 8 (9)
Hypertension (Cardiac disorders) | 2 (2) | 7 (8)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 0 (0) | 6 (8)
Supraventricular and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 3 (3) | 2 (2)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (6)
Renal/Genitourinary - Other, acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 2 (2)
Dry eye syndrome (Eye disorders) | 2 (2) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 3 (3)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Renal/Genitourinary - Other, hematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal/Genitourinary - Other, renal insufficiency (Renal and urinary disorders) | 2 (2) | 1 (1)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes